CLINICAL TRIAL: NCT03800667
Title: Vitamin C for the Prevention of UTI in Women Who Undergo Elective GYN Surgeries: a Study Protocol for a Randomized Controlled Trial
Brief Title: Vitamin C for the Prevention of UTI in Women Who Undergo Elective GYN Surgeries
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No funds
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Tony Bazi, MD, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OGY.TB.09
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Catheter-Associated Urinary Tract Infection, Ascorbic Acid
Keywords: Vitamin C, CAUTI
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Women on a vitamin C regimen (Experimental): Women who are undergoing elective gynecological surgeries and who are randomized to take 1000 mg of vitamin C for one month,
  Interventions: Drug: Ascorbic Acid 1000 MG
- Women not taking vitamin C (No Intervention): Women who are undergoing elective gynecological surgeries and who are randomized not to take any vitamin C for one month.

INTERVENTIONS:
Drug: Ascorbic Acid 1000 MG — 1000 mg ascorbic acid (Vitamin C) for 1 month post-op after an elective gynecological surgery.
  Arms: Women on a vitamin C regimen

SUMMARY:
This open-label randomized trial aims at assessing the role of Vitamin C pills in the prevention of catheter-associated urinary tract infections in women undergoing elective gynecological surgeries.

ELIGIBILITY:
Inclusion Criteria:

Non pregnant women at least 18 years of age visiting the Preadmission unit (PAU) or the OBGYN floor (7N), presenting for elective GYN surgery at the American University of Beirut Medical Center (AUBMC).

Exclusion Criteria:

* Any women with the following:

  1. Nephrolithiasis
  2. Congenital anomaly or neurogenic bladder
  3. Allergy to ascorbic acid
  4. Who require therapeutic anticoagulant medicine during the 6 weeks after surgery
  5. Surgery did involve a fistula repair or a vaginal mesh removal
  6. Positive Urinalysis in the PAU
  7. Recurrent UTI's
  8. Diabetes
  9. G6PD
  10. Hemochromatosis
  11. Renal disorders

Patients already taking Vitamin C supplementation will also be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who experienced clinically diagnosed and treated UTI. | 30 days
  Urinary tract infection is diagnosed by a positive urine culture.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Bazi, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Foxman B, Cronenwett AE, Spino C, Berger MB, Morgan DM. Cranberry juice capsules and urinary tract infection after surgery: results of a randomized trial. Am J Obstet Gynecol. 2015 Aug;213(2):194.e1-8. doi: 10.1016/j.ajog.2015.04.003. Epub 2015 Apr 13. PMID 25882919
- [Result] Ochoa-Brust GJ, Fernandez AR, Villanueva-Ruiz GJ, Velasco R, Trujillo-Hernandez B, Vasquez C. Daily intake of 100 mg ascorbic acid as urinary tract infection prophylactic agent during pregnancy. Acta Obstet Gynecol Scand. 2007;86(7):783-7. doi: 10.1080/00016340701273189. PMID 17611821
- [Result] Carlsson S, Wiklund NP, Engstrand L, Weitzberg E, Lundberg JO. Effects of pH, nitrite, and ascorbic acid on nonenzymatic nitric oxide generation and bacterial growth in urine. Nitric Oxide. 2001 Dec;5(6):580-6. doi: 10.1006/niox.2001.0371. PMID 11730365
- [Result] Trautner BW, Darouiche RO. Catheter-associated infections: pathogenesis affects prevention. Arch Intern Med. 2004 Apr 26;164(8):842-50. doi: 10.1001/archinte.164.8.842. PMID 15111369
- [Result] Barbosa-Cesnik C, Brown MB, Buxton M, Zhang L, DeBusscher J, Foxman B. Cranberry juice fails to prevent recurrent urinary tract infection: results from a randomized placebo-controlled trial. Clin Infect Dis. 2011 Jan 1;52(1):23-30. doi: 10.1093/cid/ciq073. PMID 21148516
- [Result] Hickling DR, Nitti VW. Management of recurrent urinary tract infections in healthy adult women. Rev Urol. 2013;15(2):41-8. PMID 24082842
- [Result] Wald HL, Ma A, Bratzler DW, Kramer AM. Indwelling urinary catheter use in the postoperative period: analysis of the national surgical infection prevention project data. Arch Surg. 2008 Jun;143(6):551-7. doi: 10.1001/archsurg.143.6.551. PMID 18559747